CLINICAL TRIAL: NCT01606228
Title: An Open-Label Prospective Trial to Explore the Tolerability, Safety and Efficacy of Flexibly-Dosed Paliperidone ER Among Treatment-Naïve and Newly Diagnosed Patients With Schizophrenia
Brief Title: A Trial to Explore the Tolerability, Safety and Efficacy of Paliperidone Extended Release in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Medical Director, Jan-Cil Philippines
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014452; R076477SCH3033 (Other: Janssen Pharmaceutica); PAL-PHL-MA3 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2012-05-16; First posted 2012-05-25 (Estimated); Results first posted 2012-10-22 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone ER; Treatment naive patients; Newly diagnosed patients
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone ER (Experimental)
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Type= range, unit= mg/day, number= 3 to 12, form= tablet, route= oral use. Paliperidone ER 6 mg orally administered once daily for the first five days. Thereafter, flexible dosing in a range of 3 to 12 mg/day.

SUMMARY:
The purpose of this study is to explore the tolerability, safety and efficacy of flexibly dosed paliperidone extended release (ER) among patients with schizophrenia.

DETAILED DESCRIPTION:
This is a single arm (the same intervention is given to all patients), multicenter study that aimed to explore the tolerability, safety and efficacy of flexibly dosed paliperidone extended release (ER) among Filipino patients with schizophrenia who have not taken any antipsychotics in the past, and among newly diagnosed schizophrenia patients who have not taken any antipsychotics for at least one month prior to screening. Antipsychotics are drugs that are helpful in the treatment of psychosis and have a capacity to ameliorate thought disorders. Flexible dosing allows the investigators to adjust the dosage of each patient based on the individual needs.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with schizophrenia
* Patient with Positive and Negative Syndrome Scale (PANSS) score of 80 to 120 at screening
* Patients who have not taken any antipsychotics in the past, and those were newly diagnosed with schizophrenia who have not taken any antipsychotics for at least one month prior to screening
* Patient healthy on the basis of a physical examination, laboratory examination, and vital signs
* Women must have a negative pregnancy test, and agree to practice an effective method of birth control before entry and throughout the study

Exclusion Criteria:

* Serious unstable medical condition, including known clinically relevant laboratory abnormalities
* Judged to be at high risk for adverse events, violence or self-harm
* Inability to swallow the study medication whole with the aid of water (patients may not chew, divide, dissolve, or crush the study medication)
* Biochemistry results that are out of the laboratory's normal reference range and are deemed to be clinically significant by the investigator
* Patients with a current use or known history (over the past 6 months) of substance dependence
* Positive urine drug examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 188 patients enrolled in the study which were included in the safety analysis set. The main analysis set included only 176 subjects due to 12 protocol violations. Of these 176 patients, only 73 were included in the per-protocol analysis set. For the Clinical Global Impression-Severity scores, data was collected for only 60 patients.
Groups:
- Paliperidone Extended-release (ER): Paliperidone ER 6 mg orally administered once daily for the first five days. Thereafter, flexible dosing in a range of 3 to 12 mg/day.
Period: Overall Study
Arm/Group | Paliperidone Extended-release (ER)
Started | 188
Completed | 159
Not Completed | 29
Not completed — Lost to Follow-up | 20
Not completed — Withdrawal by Subject | 3
Not completed — Non-compliant | 3
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 176
Age Continuous [Mean (Standard Deviation); unit: years] | 33.71 (9.743)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Improving 20% in Total Positive and Negative Syndrome Scale (PANSS) at Endpoint (Day 90)
Description: The PANSS is a 30-item scale (range 30-210) designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items. Higher scores indicate worsening.
Time Frame: Baseline, Day 90
Population: Per Protocol (PP) population
Measure: Number; unit: percentage of patients
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
percentage of patients | 97.73

2. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Scores at Baseline
Description: as for outcome 1
Time Frame: Baseline
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 108.25 (23.897)

3. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Scores at Day 90
Description: as for outcome 1
Time Frame: Day 90
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 48.74 (18.371)

4. Secondary Outcome: Clinical Global Impression-Severity (CGIS) Scores at Baseline
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. The rating varies from "Normal (not at all ill)" to "Extreme (among the most extremely ill patients)".
Time Frame: Baseline
Population: Per Protocol (PP) population; participants for whom CGIS data was collected.
Measure: Number; unit: participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 60
participants
  Normal | 0
  Borderline | 0
  Mild | 0
  Moderate | 11
  Marked | 33
  Severe | 14
  Extreme | 2

5. Secondary Outcome: Clinical Global Impression-Severity (CGIS) Scores at Day 90
Description: as for outcome 4
Time Frame: Day 90
Population: Per Protocol (PP) population
Measure: Number; unit: participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 60
participants
  Normal | 0
  Borderline | 31
  Mild | 20
  Moderate | 8
  Marked | 1
  Severe | 0
  Extreme | 0

6. Secondary Outcome: Personal and Social Performance (PSP) Scores at Baseline
Description: This PSP assesses the degree of a patient's dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care, and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (i, absent to vi, very severe) in each of the 4 domains. Based on the four domains there will be one total score. Patients with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; =< 30, functioning so poorly as to require intensive supervision.
Time Frame: Baseline
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 37.23 (12.675)

7. Secondary Outcome: Personal and Social Performance (PSP) Scores at Day 90
Description: as for outcome 6
Time Frame: Day 90
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 75.66 (10.451)

8. Secondary Outcome: Patient Satisfaction With Paliperidone Treatment
Description: Patients will be interviewed to assess their satisfaction with the current treatment on a 5-point scale (very good, good, reasonable, moderate or poor).
Time Frame: 90 days
Population: Per Protocol (PP) population
Measure: Number; unit: participants
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
participants
  Very good | 33
  Good | 34
  Moderate | 4
  Poor | 1
  Very poor | 1

9. Secondary Outcome: Quality of Sleep at Baseline
Description: The quality of sleep is measured by a self-administered scale in which patients indicate how well they have slept in the previous 7 days, from 0 (very badly) to 100 (very well).
Time Frame: Baseline
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 33.99 (30.091)

10. Secondary Outcome: Quality of Sleep at Day 90
Description: as for outcome 9
Time Frame: Day 90
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 86.56 (18.684)

11. Secondary Outcome: Daytime Drowsiness at Baseline
Description: The daytime drowsiness is measured by a self-administered scale in which patients indicate how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 100 (all the time).
Time Frame: Baseline
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 21.49 (22.511)

12. Secondary Outcome: Daytime Drowsiness at Day 90
Description: as for outcome 11
Time Frame: Day 90
Population: Per Protocol (PP) population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Paliperidone Extended-release (ER)
Number analyzed (Participants) | 73
scores on a scale | 11.23 (19.061)

ADVERSE EVENTS:
Arm/Group | Paliperidone Extended-release (ER)
Serious Adverse Events (participants affected / at risk) | 4/188
Other Adverse Events (participants affected / at risk) | 43/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended-release (ER) (N=188)
Schizophrenia paranoid type (Psychiatric disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Ventricular Extrasystoles (Cardiac disorders) | 1
Akathisia (Nervous system disorders) | 1
Schizophrenia (Psychiatric disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone Extended-release (ER) (N=188)
Insomnia (Psychiatric disorders) | 25
Anemia (Metabolism and nutrition disorders) | 9
Hypertension (Vascular disorders) | 3
Pyrexia (General disorders) | 3
Extra-Pyramidal Symptoms (Nervous system disorders) | 3
Akathisia (Nervous system disorders) | 3
Acute psychotic symptoms (Psychiatric disorders) | 3
Poor appetite (Metabolism and nutrition disorders) | 3
Disturbed behavior (Psychiatric disorders) | 3
Sialorrhea (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Otitis media (Infections and infestations) | 2
Restlessness (Nervous system disorders) | 2
Breast pain (General disorders) | 2
Urinary Tract Infection (Infections and infestations) | 2
Verbal assault (Social circumstances) | 2
Fungal infection (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Dizziness/Vertigo (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Colds/nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Tremors (Nervous system disorders) | 1
Dystonia (Nervous system disorders) | 1
Skin allergy (Skin and subcutaneous tissue disorders) | 1
Upward gazing (Eye disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Acute Gastroenteritis (Gastrointestinal disorders) | 1
Swelling of arm (General disorders) | 1
Sore throat (General disorders) | 1
Eczematous lesion (Skin and subcutaneous tissue disorders) | 1
External Hemorrhoid (Vascular disorders) | 1
Pharyngitis (Infections and infestations) | 1
Diabetes (Metabolism and nutrition disorders) | 1
Sprain (Musculoskeletal and connective tissue disorders) | 1
Scabies (Infections and infestations) | 1
Manic-like behavior (Psychiatric disorders) | 1
Delusions (Psychiatric disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Pulmonary Tuberculosis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No